CLINICAL TRIAL: NCT03732352
Title: Creating Metabolic Vulnerabilities in Patients with EGFR Activated Recurrent Glioblastoma by Inhibiting EGFR with Osimertinib
Brief Title: 18F-FDG PET and Osimertinib in Evaluating Glucose Utilization in Patients with EGFR Activated Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001000; NCI-2018-02010 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-10-15; First posted 2018-11-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: EGFR Gene Amplification; EGFR Gene Mutation; Glioblastoma; Recurrent Glioblastoma; Supratentorial Glioblastoma; TP53 Wt Allele
MeSH Terms: conditions — Glioblastoma | interventions — Fluorodeoxyglucose F18; osimertinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (18F-FDG PET, osimertinib) (Experimental): Within days -28 to -4, patients receive fludeoxyglucose F-18 IV and after 60 minutes undergo PET scan over 15 minutes. After 18-54 hours, patients undergo a second fludeoxyglucose F-18 PET scan. Patients then receive osimertinib PO QD on days -3 to -1 and after 24-72 hours, undergo a third fludeoxyglucose F-18 PET scan. Patients then receive osimertinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Fludeoxyglucose F-18; Drug: Osimertinib; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso
Procedure: Positron Emission Tomography — Undergo fludeoxyglucose F-18 PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET) and osimertinib works in evaluating glucose utilization in patients with EGFR activated glioblastoma. Osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. 18F-FDG PET imaging may help to detect changes in tumor glucose utilization, which may allow investigators to obtain an early read out on the impact of osimertinib on recurrent glioblastoma patients whose tumors have EGFR activation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define the test - retest variance of tumor fludeoxyglucose (FDG) uptake using double baseline 18F-FDG PET imaging (18 to 54 hours apart) in patients with EGFR activated recurrent glioblastoma.

II. After defining #1, evaluate whether osimertinib can create a statistically significant decrease in glucose utilization as determined using early, post dosing (24-72 hour) FDG-PET imaging in patients with EGFR activated recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. Safety and tolerability of osimertinib in this patient population. II. Determine clinical effect of osimertinib in this patient population, as determined by 6 months progression-free survival.

III. Correlated clinical effect of osimertinib with FDG-PET results in this patient population, to define by receiver operating characteristic (ROC) analysis a clinically meaningful decrease in glucose utilization, which correlates with the clinical effect.

IV. Evaluate pharmacokinetic (PK) in this patient population using spot PK during imaging and at set time points during the study.

OUTLINE:

Within days -28 to -4, patients receive fludeoxyglucose F-18 intravenously (IV) and after 60 minutes undergo PET scan over 15 minutes. After 18-54 hours, patients undergo a second fludeoxyglucose F-18 PET scan. Patients then receive osimertinib orally (PO) once daily (QD) on days -3 to -1 and after 24-72 hours, undergo a third fludeoxyglucose F-18 PET scan. Patients then receive osimertinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide written informed consent
* Patients must have histologically proven World Health Organization (WHO) grade IV glioblastoma who have supratentorial contrast enhancing progressive or recurrent tumor by MRI imaging following standard or experimental treatment.
* Patients must have measurable contrast enhancing disease with a measurement of at least 1 x 1 x 1 cm using MRI contrast imaging
* Patients must have recovered from severe toxicity of prior therapy. The following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any Food and Drug Administration (FDA) approved agents
  * 5 half-lives or 4 weeks, whichever is greater, from any investigational (not FDA-approved) agents
  * 4 weeks from the last treatment with bevacizumab
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent other than bevacizumab (e.g., hydroxychloroquine, etc.)
* Patient tumor sample must have evidence of EGFR activation as determined by EGFR amplification and/or EGFR mutations by fluorescent in situ hybridization (FISH) or sequencing approaches
* Patient tumor sample must not have p53 mutation

  * Note: Patients will be enrolled based on the documented EGFR/p53 status from the previous assays completed locally. If post enrollment evaluation of the archival tissue revealed that neither EGFR amplification nor EGFR mutations were present by using FISH or next generation sequencing, or mutant p53 by exon sequencing, the patients may continue their participation in the study. The investigator should discuss with patients regarding their willingness of continuation of participation in the study
* Patients must have a Karnofsky performance status (KPS) >= 60
* Patients must have a life expectancy >= 12 weeks
* Patients must be able to swallow medication by mouth
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of osimertinib administration
* Provision of informed consent for genetic research

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study or previous treatment with osimertinib
* Prior exposure to EGFR targeted therapy
* Currently receiving any other investigational agents
* Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 weeks prior)
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2, prior platinum-therapy? related neuropathy
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator?s opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 msec obtained from an electrocardiogram (ECG), using the screening clinic ECG machine derived QTc value
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Absolute neutrophil count < 1.5 x 10^9/L
* Platelet count < 100 x 10^9/L
* Hemoglobin < 90 g/L
* Alanine aminotransferase > 2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
* Aspartate aminotransferase > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
* Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert?s syndrome (unconjugated hyperbilirubinemia) or liver metastases
* Serum creatinine > 1.5 times ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by Cockcroft and Gault equation)?confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
* History of hypersensitivity active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Intrapatient variance of tumor fludeoxyglucose F-18 (FDG) uptake as determined by a double baseline FDG positron emission tomography (PET) prior to osimertinib exposure | At baseline
  Test-retest variances in FDG uptake will be estimated considering the variance of sample specific differences between first and second PET scans. This variance component will be estimated using a Bayesian conjugate analysis of Gaussian variates. Model adequacy diagnostics will compare predictive distributions to the observed data via posterior predictive assessment. Bayesian (95%) high posterior density intervals, and Bayesian posterior means will be used as the basis for statistical inference.
Change in FDG uptake in tumor after short course exposure to osimertinib | Baseline to day -1
  In order to estimate the difference in FDG tumor uptake between pre and post exposure to osimertinib, a simple change model will be considered, comparing the mean baseline uptake with the mean uptake, after treatment. A formal test for difference in mean will be based on a paired T statistic for difference in mean. 95% confidence intervals will be used to quantify uncertainty in estimation.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 2 years
  All events will be recorded from the time a subject has signed the Informed Consent Form. AE analyses will include only treatment emergent adverse events. Specifically, following quantities will be estimated: incidence (number [no.] of patients) and frequency (no. of events) overall and broken down by System Organ Classification and incidence (no. of patients) and frequency (no. of events) broken down by severity.
Percentage of participants surviving 6 months from the start of study treatment without progression of disease determined by progression free survival (PFS) according to Response Assessment in Neuro-oncology criteria | From the date of study treatment initiation to the date of the first documented progression or to death due to any cause, assessed up to 6 months
  Will be based on the sampling distribution of a simple binomial proportion. Additionally, descriptive data will be provided for the duration of PFS as a Kaplan-Meier curve.
Correlation between the reduction in glucose uptake and 6 months PFS | Up to 2 years
  Reduction in glucose uptake will be correlated with clinical outcome-- 6 months PFS, receiver operating characteristic curve (ROC) analyses of simple thresholding strategies will be performed using leave one out cross validation.
Concentrations of osimertinib and metabolites AZ5104 and AZ7550 in post-dosing plasma samples. | At the end of Cycle 1 (each cycle is 28 days).
  PK concentration data will be summarized using appropriate summary statistics

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cloughesy, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States